CLINICAL TRIAL: NCT00992966
Title: Vibration Response Imaging (VRI) in Children With Acute Respiratory Symptoms.
Status: Suspended | Type: Observational
Why Stopped: Study initiation has been delayed due to Sponsor decision
Sponsor: Deep Breeze (Industry)
Responsible Party: Merav Gat / VP Clinical Affairs, Deep Breeze
Other Study IDs: DB048
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-08

CONDITIONS: Pneumonia
Keywords: to acquire database of pneumonia cases in children
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The VRI device may provide a complementary diagnostic tool for lung examination and aid the physician in determining whether a chest x-ray should be performed.

DETAILED DESCRIPTION:
This study is a prospective, single center study to determine the value of VRI images as an aid in determining whether a chest x ray is necessary to evaluate children presenting with acute respiratory complaints.

Study participants will be children, selected from the Emergency Department (ED), who were designated to undergo a PA and Left Lateral CXR because of acute respiratory complaints such as a new respiratory condition, acute cough, onset of shortness of breath, or fever.

Patients who meet the study inclusion and exclusion criteria will be enrolled and will be recorded by the VRI device.

A technician will perform a CXR on the enrolled patients. The CXR and the VRI will be performed on the same day within 6 hours of each other.

VRI readers, who are blinded to the patient's CXR, history, and physical exam, will evaluate the VRI recording. The VRI reader will review the VRI images and, using the lexicon of images supplied by Deep Breeze, determine whether the VRI is normal or abnormal.

Certified radiologists will review the patient's CXR and will determine whether the CXR is normal or abnormal based solely on the CXR.

The VRI readers determination of normal or abnormal for each subject will be compared to the radiologists determination of normal or abnormal CXR for each subject.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's parent or legal guardian, is able and willing to read the Informed Consent, understands the Informed Consent, and provides written Informed Consent for the subject; if the minor child is in fact able to give consent, the minor's consent must be obtained in addition to the consent of the minor's legal guardian.
2. Boy or girl in the age range of 3-18 years.
3. Patient presented with acute respiratory complaints, acute cough, onset of shortness of breath, or fever.
4. Patient referred by ED physician and presented for CXR.

Exclusion Criteria:

1. Body habitus or skin condition that might prevent the placement of the sound sensors on the back (e.g. severe scoliosis, kyphosis, chest wall deformation, skin lesion on the back or compression fracture);
2. Potentially contagious skin lesion on the back;
3. Subject has had lung surgery;
4. Subject was prescribed the CXR for monitoring or follow up of a lung condition that pre-existed the current, acute symptoms.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total number of 80 patients in the age range of 3-18 and consisting of both boys and girls, preferably in an equal distribution
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Liora Kornreich, M.D, Principal Investigator — Shnider medical center; Liora Kornreich, Professor, Principal Investigator — Shnider medical center